CLINICAL TRIAL: NCT03801486
Title: The Effects of Incorporating Sprouted and Non-sprouted Chickpea Flour in Pasta Products Analyzed in Vivo Flow-mediated Dilation
Brief Title: Effects of Incorporating Sprouted and Non-sprouted Chickpea Flour in Pasta Products Analyzed in Vivo Flow-mediated Dilation
Status: Completed | Type: Observational
Sponsor: Montclair State University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-16-133
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2019-01

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental (SCF40): At the experimental data collection visits participants consumed 255g of pasta made with 40% sprouted chickpea flour and 60% semolina flour (SCF40) with butter.
  Interventions: Other: Experimental: Sprouted Chickpea Flour
- Control (SEM100): At the control data collection visits participants consumed 255g of pasta made with 100% semolina flour (SEM100) with butter.
  Interventions: Other: Control: Semolina Flour

INTERVENTIONS:
Other: Experimental: Sprouted Chickpea Flour — 255g of pasta with 40% sprouted chickpea flour and 60% semolina flour (SCF40) with butter.
  Other Names: SCF40
  Groups: Experimental (SCF40)
Other: Control: Semolina Flour — 255g of pasta with 100% semolina flour (SEM100) with butter.
  Other Names: SEM100
  Groups: Control (SEM100)

SUMMARY:
The investigators examined the effects on post-digestion brachial artery flow mediated dilation (FMD) and in vitro antioxidant capacity of 40% semolina flour replacement with sprouted chickpea flour.

DETAILED DESCRIPTION:
The purpose of the current study was to examine in-vitro and in-vivo effects of replacing 40% of semolina flour with sprouted chickpea flour for the use in pasta. Antioxidant capacity in-vitro was measured by Trolox Equivalent Antioxidant Capacity. Brachial artery flow-mediated dilation, a test of in-vivo endothelial function, was performed for assessment of effects on post-digestion endothelial function. The investigators hypothesized that FMD would be higher after consuming 40% of semolina flour with sprouted chickpea flour pasta vs. 100% of semolina flour pasta.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult

Exclusion Criteria:

* have diabetes mellitus, kidney disease, a history of cancer, cardiac issues, pulmonary disease, history of a stroke, obesity (for most people this means a body mass index greater than 30), or any life threatening chronic conditions.
* food allergies relevant to wheat, gluten, chickpea, and pasta sauce.
* are currently being treated for infectious mononucleosis, hepatitis, pneumonia, or other infectious diseases.
* are unable or unwilling to refrain from recreational drug (marijuana, cocaine, etc.) or alcohol use during the 24 hours prior to your exercise session.
* use nicotine products, or non-contraceptive hormonal therapy (birth control is okay).
* are pregnant or trying to become pregnant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Post-digestion flow mediated dilation | Two hours following meal
  Post meal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruno JA, Feldman CH, Konas DW, Kerrihard AL, Matthews EL. Incorporating sprouted chickpea flour in pasta increases brachial artery flow-mediated dilation. Physiol Int. 2019 Sep 1;106(3):207-212. doi: 10.1556/2060.106.2019.21. Epub 2019 Sep 30. PMID 31564118